CLINICAL TRIAL: NCT01640561
Title: Enhancing Ugandan HIV-Affected Child Development With Caregiver Training
Acronym: MISC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Michigan State University (Other); Global Health Uganda LTD (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Judith Bass, Associate Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JHU-MSU-UGANDA-2012; R01HD070723-01 (NIH)
Record Dates: First submitted 2012-07-10; First posted 2012-07-13 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: HIV
Keywords: HIV affected; Child Neurodevelopment; Low and Middle Income Country

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MISC (Experimental): The Mediational Interventions for Sensitizing Caregivers (MISC) model developed by Professor Pnina Klein (consultant) has been used to enhance the development of children throughout the developing world, with the support of such international aid agencies as the World Health Organization (WHO), UNICEF, Norwegian Agency for Development Cooperation (NORAD), and Redd Barna (Norway).
  Interventions: Behavioral: MISC
- Enhanced Treatment as Usual (Active Comparator)
  Interventions: Behavioral: UCOBAC

INTERVENTIONS:
Behavioral: MISC — The Mediational Interventions for Sensitizing Caregivers
  Arms: MISC
Behavioral: UCOBAC — This nutrition/healthcare curriculum for children in poverty and affected by HIV was developed by a non-governmental organization (NGO) operating in Uganda called Uganda Community Based Association for Child Welfare (UCOBAC) with support from UNICEF.
  Arms: Enhanced Treatment as Usual

SUMMARY:
Early childhood (up to age 5 yrs) is a period of dramatic change in the cognitive, emotional, social, and behavioral domains; children continuously progress by observing and interacting with the world around them. In the face of economic instability and nutritional, medical and educational deprivation, HIV-affected very young children are the most vulnerable HIV subgroup globally because their families are often the most vulnerable, with little margin for sustaining a favorable developmental milieu for the child. Through strategic caregiver interventions during this sensitive period of child neurodevelopment, our study findings have the potential for positively re-directing the developmental trajectories of tens of millions of HIV-affected children globally.

DETAILED DESCRIPTION:
Background. Children up to the age of 5 years affected by HIV are the most vulnerable subgroup of HIV populations globally, especially in low-resource areas. This is because of the strategic, volatile, and vulnerable nature of this highly sensitive period of child development. Mediational intervention for sensitizing caregivers (MISC) has a structured training program to enable caregivers to improve their children's cognitive and social development during everyday casual interactions in the home. In our preliminary National Institute of Mental Health (NIMH) R34 findings, Ugandan HIV children of caregivers receiving MISC training biweekly for a year showed significantly greater gains on the Mullen Early Learning Scales Composite of g fluid intelligence, when compared to children whose caregivers received a standard health/nutrition education intervention (treatment as usual or TAU). The MISC caregivers were also significantly less depressed, and their child mortality that year was significantly lower. Intervention Method. The plan was to recruit approximately 100 Ugandan HIV-positive preschool and 200 HIV orphan caregiver/child dyads will be enlisted from Tororo District. These dyads will be randomly assigned by village clusters to either biweekly MISC or health/nutrition education TAU intervention for one year. Child Outcomes are the child development gains on the Mullen, the Early Childhood Vigilance Test (ECVT) of attention, and the Color-Object Association Test (COAT) of memory, the Behavior Rating Inventory of Executive Functioning - Preschool (BRIEF-P), and the caregiver administered version of the Achenbach Child Behavior Checklist (CBCL). Caregiver Outcomes include an array of emotional wellbeing (EWB) and daily functioning measures validated during the initial qualitative study phase. Study Aim 1 will evaluate if MISC significantly enhances child outcomes when compared to controls for both HIV-positive and orphan children when assessed from baseline to 6, 12 and 24 months. Study Aim 2 will evaluate if MISC significantly enhances caregiver EWB and daily functioning outcomes. To better understand the mechanisms of MISC-enhanced child development, a Secondary Aim is to evaluate the mediating effect of improved caregiver EWB outcomes on corresponding child development gains, and the modifying effects of caregiver HIV illness and functioning on child outcomes. The Overall Impact comes from establishing the feasibility, acceptability, and effectiveness of MISC for HIV orphans and vulnerable children (OVC) and their caregivers in low resource settings; the sustainability of MISC in low resource settings since it is not dependent on published materials or outside resources; the complementary dual impact of significant psychotherapeutic benefit for the caregiver, especially mothers struggling with HIV disease. MISC will also reduce HIV child mortality because in our initial R34 findings, MISC heightened maternal bonding, sensitivity to serious illness, and the prompter seeking of medical care. It also can improve treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* Child age 1 through 5 years of age. If more than one child in a household qualifies, they will all be included.
* HIV-infected or HIV-affected child who is an orphan (loss of one or both biological parents to HIV). In either case, child must have been born to a confirmed HIV-positive mother.
* Principal caregiver of the eligible study child is able and willing to participate in a regular treatment program. The minimum agreed to participation requirement is biweekly for entire year alternating between home and office, including regular visits at 6-month intervals to the study clinic to complete lab and developmental assessments for the study child.

Exclusion Criteria:

* Child illness or injury-based central nervous system (CNS) insults which are likely to overshadow the neurocognitive benefits of sensitive-period caregiver interventions.
* Medical history of serious birth complications, severe malnutrition, bacterial meningitis, encephalitis, cerebral malaria, or other known brain injury or disorder requiring hospitalization or continued evidence of seizure or other neurological disability.
* Current enrollment or plans for enrollment in P1 (1st grade) level of school during the first 8 months of the yearlong intervention period. Having the study child in school all day precludes necessary caregiver access to child for adequate opportunity to implement MISC training with that child. We do not expect this criterion to be problematic given that age 6 is generally the age for P1.
* Primary caregiver cannot respond to MISC or TAU intervention because of mental illness or disability.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 341 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in Child Neurodevelopment post treatment | 12 month follow up
  Mullen Scales of Early Learning

SECONDARY OUTCOMES:
Change in caregiver mental health and well being | 6-, 12-, and 24-month follow ups
  Caregiver mental health will be assessed using the Hopkins Symptom Checklist (HSCL)
Midterm change in child neurodevelopment | 6-month follow up
  Mullen Scales of Early Learning, Early Childhood Vigilance Test (ECVT). Behavior Rating Inventory of Executive Function-Preschool (BRIEF-P).
Change in long term child neurodevelopment outcomes | 24-month follow ups
  Mullen Scales of Early Learning, Early Childhood Vigilance Test (ECVT). Behavior Rating Inventory of Executive Function-Preschool (BRIEF-P).
Change in child physical health and well-being | 6-, 12-, 24-month follow ups
  Measures of child growth (height and weight) and assessments of medical visits

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boivin, PhD, Principal Investigator — Michigan State University; Judy Bass, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Global Health Uganda, Tororo, Uganda

REFERENCES:
- [Background] Boivin MJ, Nakasujja N, Familiar-Lopez I, Murray SM, Sikorskii A, Awadu J, Shohet C, Givon D, Ruisenor-Escudero H, Schut EE, Opoka RO, Bass JK. Effect of Caregiver Training on the Neurodevelopment of HIV-Exposed Uninfected Children and Caregiver Mental Health: A Ugandan Cluster-Randomized Controlled Trial. J Dev Behav Pediatr. 2017 Nov/Dec;38(9):753-764. doi: 10.1097/DBP.0000000000000510. PMID 28991146
- [Background] Bass JK, Opoka R, Familiar I, Nakasujja N, Sikorskii A, Awadu J, Givon D, Shohet C, Murray SM, Augustinavicius J, Mendelson T, Boivin M. Randomized controlled trial of caregiver training for HIV-infected child neurodevelopment and caregiver well being. AIDS. 2017 Aug 24;31(13):1877-1883. doi: 10.1097/QAD.0000000000001563. PMID 28609401
- [Background] Murray SM, Familiar I, Nakasujja N, Winch PJ, Gallo JJ, Opoka R, Caesar JO, Boivin MJ, Bass JK. Caregiver mental health and HIV-infected child wellness: perspectives from Ugandan caregivers. AIDS Care. 2017 Jun;29(6):793-799. doi: 10.1080/09540121.2016.1263722. Epub 2016 Dec 13. PMID 27951734
- [Background] Familiar I, Nakasujja N, Bass J, Sikorskii A, Murray S, Ruisenor-Escudero H, Bangirana P, Opoka R, Boivin MJ. Caregivers' depressive symptoms and parent-report of child executive function among young children in Uganda. Learn Individ Differ. 2016 Feb;46:17-24. doi: 10.1016/j.lindif.2015.01.012. Epub 2015 Jan 30. PMID 27175052
- [Background] Familiar I, Murray S, Ruisenor-Escudero H, Sikorskii A, Nakasujja N, Boivin MJ, Opoka R, Bass JK. Socio-demographic correlates of depression and anxiety among female caregivers living with HIV in rural Uganda. AIDS Care. 2016 Dec;28(12):1541-1545. doi: 10.1080/09540121.2016.1191609. Epub 2016 May 30. PMID 27240825
- [Background] Bass JK, Nakasujja N, Familiar-Lopez I, Sikorskii A, Murray SM, Opoka R, Augustinavicius J, Boivin MJ. Association of caregiver quality of care with neurocognitive outcomes in HIV-affected children aged 2-5 years in Uganda. AIDS Care. 2016;28 Suppl 1(sup1):76-83. doi: 10.1080/09540121.2016.1146215. Epub 2016 Feb 17. PMID 26888568
- [Background] Seffren V, Familiar I, Murray SM, Augustinavicius J, Boivin MJ, Nakasujja N, Opoka R, Bass J. Association between coping strategies, social support, and depression and anxiety symptoms among rural Ugandan women living with HIV/AIDS. AIDS Care. 2018 Jul;30(7):888-895. doi: 10.1080/09540121.2018.1441969. Epub 2018 Feb 22. PMID 29471677
- [Derived] Boivin MJ, Augustinavicius JL, Familiar-Lopez I, Murray SM, Sikorskii A, Awadu J, Nakasujja N, Bass JK. Early Childhood Development Caregiver Training and Neurocognition of HIV-Exposed Ugandan Siblings. J Dev Behav Pediatr. 2020 Apr;41(3):221-229. doi: 10.1097/DBP.0000000000000753. PMID 31800526
- [Derived] Ruisenor-Escudero H, Sikorskii A, Familiar-Lopez I, Persaud D, Ziemniak C, Nakasujja N, Opoka R, Boivin M. Neruodevelopmental Outcomes in Preschool Children Living With HIV-1 Subtypes A and D in Uganda. Pediatr Infect Dis J. 2018 Dec;37(12):e298-e303. doi: 10.1097/INF.0000000000002097. PMID 29746376